CLINICAL TRIAL: NCT00005483
Title: Plasma Homocysteine Distribution in the United States
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4970; R01HL052630 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hyperhomocysteinemia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hyperhomocysteinemia

SUMMARY:
To describe the distribution of homocysteine and prevalence of hyperhomocysteinemia with emphasis on race, sex and age. To determine the extent to which hyperhomocysteinemia is associated with status of folate and vitamin B12. Finally, to describe the relationships between prevalence of hyperhomocysteinemia and prevalence of cardiovascular disease and assess the importance of this risk factor as a cause of vascular disease among US adults. The study was renewed for one year to investigate normal homocysteine concentrations among children and to identify nutritional and non-nutritional determinants of total homocysteine concentrations in children.

DETAILED DESCRIPTION:
BACKGROUND:

Hyperhomocysteinemia, a condition of elevated plasma homocysteine concentrations resulting from impaired sulfur amino acid metabolism, may be a powerful risk factor for occlusive vascular disease. However, little is known about the distribution of hyperhomocysteinemia in the general population. Furthermore, inadequate nutritional status might be a strong determinant of hyperhomocysteinemia, but its importance at a population level (as measured by the prevalence of hyperhomocysteinemia associated with inadequate nutrition) has received little study. Finally, levels of homocysteine associated with elevated risk of vascular disease have not been clearly established.

DESIGN NARRATIVE:

Using previously collected plasma samples, studies were conducted on the distribution of homocysteine and prevalence of hyperhomocysteinemia with emphasis on race, sex and age. Investigations were undertaken on the extent of the relationship of hyperhomocysteinemia to folate and vitamin B12. Finally, the relationships were described between prevalence of hyperhomocysteinemia and prevalence of cardiovascular disease and the importance of this risk factor as a cause of vascular disease among US adults was assessed..

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-12; Study Completion 1999-07

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Selhub — Tufts University

REFERENCES:
- [Background] Selhub J, Jacques PF, Rosenberg IH, Rogers G, Bowman BA, Gunter EW, Wright JD, Johnson CL. Serum total homocysteine concentrations in the third National Health and Nutrition Examination Survey (1991-1994): population reference ranges and contribution of vitamin status to high serum concentrations. Ann Intern Med. 1999 Sep 7;131(5):331-9. doi: 10.7326/0003-4819-131-5-199909070-00003. PMID 10475885
- [Background] Jacques PF, Rosenberg IH, Rogers G, Selhub J, Bowman BA, Gunter EW, Wright JD, Johnson CL. Serum total homocysteine concentrations in adolescent and adult Americans: results from the third National Health and Nutrition Examination Survey. Am J Clin Nutr. 1999 Mar;69(3):482-9. doi: 10.1093/ajcn/69.3.482. PMID 10075334